CLINICAL TRIAL: NCT05967559
Title: Effect Of The Online Flipped Learning Model on Students' Achievement, Critical Thinking Dispositions, and Self-Directed Learning Skills
Brief Title: Online Flipped Learning in Nursing Student
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Erden, Principal Investigator Dr., Namik Kemal University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: DeRDEN
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy Effect
Keywords: academic achievement; chemotherapy; critical thinking; online learning; nursing students; active learning

STUDY DESIGN:
Intervention Model Description: The students who were informed about the research, and after obtaining their individual consent, the Chemotherapy Symptom Management Knowledge Test , the Marmara Critical Thinking Dispositions Scale , and the Self-Directed Learning Skills Scale were administered using an online questionnaire. Chemotherapy symptom management training was conducted online for six weeks, one hour per week, for experiment and control groups. The research began with the control group to minimize the interaction between the students in the experiment and control groups. Then the experiment group practices were carried out after the control group's program was completed.
Who Masked: Participant
Masking Description: The aim of the research was to reduce the bias by using a single-blind technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): The experimental group received online flipped learning training for six weeks.
  Interventions: Other: Online Flipped Learning Group
- Control groups (Other): The control group received traditional learning training for 6 weeks.
  Interventions: Other: Traditional learning Group

INTERVENTIONS:
Other: Online Flipped Learning Group — The experimental group is the group that receives online flipped learning training.
  Arms: Experiment group
Other: Traditional learning Group — The control group is the group that received traditional learning training.
  Arms: Control groups

SUMMARY:
Cancer is one of the major health problems facing Turkey and the world. One of the methods used to treat cancer is chemotherapy. During this treatment period, some side effects may develop in patients. These developing symptoms can be managed with effective nursing interventions, which in turn can increase the patient's quality of life. Managing these symptoms is among the responsibilities of the nurse. The nurses' ability to effectively manage the side effects of chemotherapy depends on gaining specific knowledge, attitudes, and skills during their vocational training and the development of problem-solving and critical thinking. The research was carried out to examine the effect of chemotherapy symptom management education based on the online flipped learning model on the achievement, critical thinking, and self-directed learning of nursing students.

DETAILED DESCRIPTION:
Background: The online flipped learning method is an innovative learning approach that helps develop critical thinking and self-directed learning skills and increases students' interest in the course Aim: The research was carried out to examine the effect of chemotherapy symptom management education based on the online flipped learning model on the achievement, critical thinking, and self-directed learning of nursing students.

Methods: This research is a randomized controlled trial. The sample consisted of 68 students divided into experiment and control groups. The training program based on traditional learning was applied to the control group, online flipped learning was applied to the experiment group, and each group received training on chemotherapy symptom management for one hour per week for six weeks. The researchers evaluated the results by applying the Chemotherapy Symptom Management Knowledge Test (CSMKT), the Marmara Critical Thinking Dispositions Scale (MCTDS), and the Self-Directed Learning Skills Scale (SDLSS) to the control and experiment groups before, right after the training, and one month after the training.

ELIGIBILITY:
Inclusion Criteria:

* Second-year students who took the course basics of nursing, internal medicine nursing, physiology, pathology, and computer courses and were able to actively use the computer and voluntarily participated in the research were included.

Exclusion Criteria:

* Students in other classes
* Those who did not volunteer to participate in the study

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Chemotherapy Symptom Management Knowledge Test (CSMKT) | 1 month
  The Chemotherapy Symptom Management Knowledge Test (CSMKT) was developed by the researchers to evaluate the impact of chemotherapy symptom management training based on the online flipped learning model. The measurement tool was presented to the expert opinion. Necessary corrections were made in accordance with the views of the experts and validity and reliability analyzes were carried. The test consists of 25 questions with a total of five options.The minimum score that can be attainable from the scale is 0, and the maximum score is 100. As the total score increases, the academic success of the student increases.

SECONDARY OUTCOMES:
Marmara Critical Thinking Dispositions Scale (MCTDS) | 1 month
  The MCTDS was developed by Özgenel and Çetin (2018). The scale includes 28 items and six subdimensions: reasoning (six items), reaching judgment (six items), searching for evidence (four items), searching for the truth (four items), open-mindedness (four items), and systematicity (four items). It is a five-point Likert-type scale (5 = Always, 1 = Never). There are no reverse-scored items in the scale. The minimum score that can be attainable from the scale is 28, and the maximum score is 140. The Cronbach's alpha internal consistency coefficient of the scale was determined as α = 0.91 As the total score increases, the student's critical thinking dispositions increases.
Self-Directed Learning Skills Scale (SDLSS) | 1 month
  The SDLLS was developed by Aşkın Tekkol and Demirel (2018). The scale includes 21 items and four subdimensions: motivation (seven items), self-control (five items), self-monitoring (five items), and self-confidence (four items). It is a five-point Likert-type scale (1 = Always, 5 = Never). There are no reverse-scored items in the scale. While the minimum score of the scale is 21, the maximum score is 105. The overall reliability, the Cronbach's alpha internal consistency coefficient, was determined as α = 0.89. As the total score increases, the student's self-directed learning skills increases.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Erden, PhD., Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdağ Namık Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No